CLINICAL TRIAL: NCT04307329
Title: Monalizumab and Trastuzumab In Metastatic HER2-pOSitive breAst Cancer: MIMOSA-trial
Acronym: MIMOSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N19MIM
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: HER2 positive; Metastatic disease; Accessible lesion for study biopsies; Min 1, max 3 lines palliative treatment
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — monalizumab; Trastuzumab

STUDY DESIGN:
Intervention Model Description: Simon's two-stage minimax design
Masking Description: Two cohorts; high TILs (≥ 5%) and low (< 5%) TILs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monalizumab + trastuzumab - low TILs (<5%) (Experimental): trastuzumab 4 mg/kg and monalizumab 750 mg every two weeks.
  Interventions: Biological: Monalizumab; Biological: Trastuzumab
- Monalizumab + trastuzumab - high TILs (>=5%) (Experimental): trastuzumab 4 mg/kg and monalizumab 750 mg every two weeks.
  Interventions: Biological: Monalizumab; Biological: Trastuzumab

INTERVENTIONS:
Biological: Monalizumab — Monalizumab 750 mg every two weeks
Biological: Trastuzumab — Trastuzumab 4 mg/kg every two weeks

SUMMARY:
In this phase II clinical trial the efficacy of the combination of monalizumab and trastuzumab is assessed in patients with metastatic or locally incurable HER2-positive breast cancer

DETAILED DESCRIPTION:
In this phase II clinical trial with an explorative nature, the efficacy of the combination of monalizumab and trastuzumab is assessed in patients with metastatic or locally incurable HER2-positive breast cancer. Clinical efficacy will be assessed in patients with high stromal tumor-infiltrating lymphocytes (sTILs) or low sTILs in two separate cohorts (higher or equal to 5% versus lower than 5%). Since the combination of monalizumab and trastuzumab has not been administered before, dose limiting toxicities (DLTs) will be monitored throughout the trial using the Pocock-type boundary rules for continuous monitoring of toxicity in phase II trials.

In the first stage, 11 patients will be accrued per cohort. If there are 1 or fewer responses in these 11 patients, the study will be stopped. Otherwise, 8 additional patients will be accrued for a total of 19 patients.

The study will start with two cohorts (sTILs high and sTILs low), a total of 22 (2x11) patients will be included in the first stage. Dependent on the interim analysis (continuation of no cohorts, 1 or 2 cohorts), a maximum of 38 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

without SISH amplification) breast cancer. HER2-positivity must have been assessed on a metastatic lesion.

* Histological or cytological confirmed locally incurable or metastatic disease
* Accessible lesion for study biopsies.
* Administration of at least one line of palliative treatment with documented progression and a maximum of three lines of palliative chemotherapy in combination with HER2 targeting agents (TDM-1 is considered one line of palliative treatment). Trastuzumab in combination with endocrine treatment is not defined as one line of treatment.
* Documented progression during previous trastuzumab-based therapy
* Measurable disease according to RECIST1.1 (at least one target lesion)
* Left ventricular ejection fraction of 50% or higher
* WHO performance status of 0 or 1
* No signs of a visceral crisis
* Signed written informed consent - Subjects with brain metastases are eligible if they have been treated, asymptomatic and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks prior to study registration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration

Exclusion Criteria:

* uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris
* known leptomeningeal disease localization
* history of having received other anticancer therapies within 2 weeks of start of the study drug
* history of immunodeficiency, autoimmune disease, conditions requiring innmunosuppression (>10 mg daily prednisone equivalents) or chronic infections. Subjects with vitiligo, diabetes mellitus type I on a stable insulin regimen, psoriasis not requiring systemic treatment or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections will not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement, Sjogren's syndrome or conditions not expected to recur in the absence of an external trigger will not be excluded from the study. Adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoinnmune disease
* prior treatment with immune checkpoint blockade or other forms of imnnunotherapy, such as but not limited to: anti-PD-(L)1, anti-PD-L2, anti-CTLA-4, anti-GITR or CD137/0X40 agonists
* prior treatment with HER2-based vaccines
* live vaccine within two weeks prior to start of the study, at any time during the study or within 5 months following the last dose of monalizumab. Inactivated vaccines, such as the seasonal flu vaccination, are allowed
* history of clinically significant or uncontrolled cardiac disease, including congestive heart failure (New York Heart Association functional classification .3), angina, myocardial infarction within 12 months prior to study treatment or ventricular arrhythmia.
* active other cancer
* positive test for hepatitis B surface virus surface antigen (HBsAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* allogeneic stem cell or organ transplantation, HIV or active tuberculosis
* history of uncontrolled serious medical or psychiatric illness
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* current pregnancy or breastfeeding. Women of childbearing potential (WOCBP) must use adequate contraceptive protection. WOCBP must have a negative serum or urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2024-03-23 (Actual)

PRIMARY OUTCOMES:
Response | to be assessed up to 120 months
  number of patients with partial response or complete response according to RECIST1.1

SECONDARY OUTCOMES:
Clinical Benefit | to be assessed every 8 weeks up to 120 months
  number of patients with complete response, partial response or stable disease for more than 24 weeks according to RECIST1.1
Progression Free Survival | assessed up to 120 months
  From date of registration until date of first documented progression or date of death, which ever comes first
Overall survival | assessed up to 120 months
  From date of registration until date of death
Toxicity; incidence of toxicity | assessed every 2 weeks until 30 days after last study treatment
  Adverse events will be graded according to NCI Common Toxicity Criteria version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Kok, MD, Principal Investigator — NKI-AvL
Locations (1):
- NKI-AVL, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
to be detemined